CLINICAL TRIAL: NCT04005027
Title: Exercise Induced Inter-individual Responses in QT Interval Duration and Dispersion During and Following Intermittent and Continuous Graded Exercise Tests in Young Male Football Players
Brief Title: Exercise Induced QT Interval Changes in Response to Intermittent and Continuous Graded Exercise Tests
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is currently suspended due to ongoing risks of infection, and unknown risks to participants as a consequence of the Covid-19 pandemic.
Sponsor: University of Sunderland (Other)
Collaborators: Sheffield Hallam University (Other); Newcastle University (Other); Teesside University (Other)
Responsible Party: Principal Investigator, Will Evans, Principle Investigator, University of Sunderland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LQT004291
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Qt Interval, Variation in
Keywords: QT interval; Intermittent Exercise; Continuous Exercise; Cardiac; Electrocardiogram

STUDY DESIGN:
Intervention Model Description: The investigators will use a replicated randomised repeated measures crossover design in which the participants will be randomised to different sequences of four experimental conditions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent graded exercise (INT) (Experimental): The intermittent graded exercise test (INT) increase treadmill speed incrementally using three minute stage duration on a motorised treadmill. However, the speed within each three minute exercise bout will vary every 30 s between the target speed, and a complete pause for 30 s. The acceleration of the treadmill belt will be set to its maximum capability.
  Interventions: Other: Intermittent graded exercise test
- Continuous graded exercise (CONT) (Active Comparator): The continuous graded exercise test (CONT) will increase treadmill speed incrementally using three minute stage duration on a motorised treadmill
  Interventions: Other: Intermittent graded exercise test

INTERVENTIONS:
Other: Intermittent graded exercise test — Participants will run on a treadmill until volitional exhaustion. The speed of the treadmill belt will increase incrementally every 3 minutes. Within each 3 minute stage the speed will vary between the target speed and a complete pause (e.g target speed = 8 km/hr)

SUMMARY:
Long QT syndrome (LQTS) is an inherited heart defect where the heart takes longer to recover between beats. LQTS is a known condition predisposing young footballers to sudden cardiac death (SDC). The existence of LQTS can be established by measuring the QT interval in an electrocardiogram (ECG). Currently pre-participation cardiac screening is performed in young athletes but players may only be screened at 16 years old using only a resting ECG, and a medical check including a questionnaire on family and medical history. However, the sensitivity and specificity of the screening to investigate underlying causes of SCD could be improved with the addition of an exercise stress test or cardiopulmonary exercise test (CPET). Certain abnormalities in the heart may only become apparent when the heart has been stressed (e.g. via exercise). This is particularly important as in young athletes these abnormal rhythms manifest during rest and recovery rather than at peak exercise. The CPET measures changes in the ECG in response to exercise that increases in intensity in a continuous manner until the participant cannot exercise any long. However, football is characterised by high- intensity bouts of exercise interspersed with low-intensity bouts or pauses. Therefore, the continuous test does not reflect the movement patterns of football and may not stress the cardiovascular system in a similar manner. To address this, intermittent graded exercise tests have been developed to reflect the intermittent movement pattern. As yet there is limited evidence on whether there are any differences in ECG changes during intermittent exercise. Specifically, it is not clear how an intermittent movement pattern might affect the QT interval.

DETAILED DESCRIPTION:
Long QT syndrome (LQTS) is an ion channelopathy which occurs in approximately 1 in every 2500 individuals. Symptoms include; syncope, seizures and sudden cardiac death (SCD). LQTS's genetic defects culminate in delayed cardiac repolarization identified on a 12 lead electrocardiogram (ECG) as a prolonged QT interval. Due to the dynamic nature of channelopathies, some abnormalities could be missed with a resting ECG alone. In young athletes cardiac arrhythmia's predisposing athletes to SCD do not usually occur at peak exercise but during warm-up, recovery or periods of reduced exercise intensity (e.g. rest phases in football games). Environments causing increase in body temperature, heat rate, and autonomic status should therefore be included in the assessment of risk of SCD. Whilst the use of cardiopulmonary exercise testing (CPET) is commonplace, the use of such an exercise test is often performed using a continuous ramp or step procedure (e.g Bruce protocol). However, during games play such as football, movements are not continuous but intermittent characterised by rest phases and lower intensity periods of exercise. The primary aim of this study is to assess the duration and dispersion of the QT interval during and immediately following the performance of a continuous (CONT), and an intermittent (INT) maximal graded exercise test in a group of young (< 16-18 yr) semi-professional soccer players. It is anticipated that the INT graded exercise test will induce greater inter-individual variability in the QT interval compared to the CONT trial.

The investigators aim to recruit approximately 50 players from Sunderland Foundation of Light regional training centre (RTC) with a minimum sample size of 24. We will use a replicated randomised repeated measures crossover design in which the participants will be randomised to different sequences of four experimental conditions; two continuous graded exercise tests, and two intermittent graded exercise tests, randomised using a Latin square counterbalanced design. Participants will be required to perform all four exercise conditions at approximately the same time of day (± 1 h) to control for within-athlete variation. Each exercise condition will be separated by at least 72 h with all testing sessions complete within a 2-4 week period. The following constraints will be placed on the participants to improve the strength of the study design:

* Avoid strenuous physical activity for 48-72 h prior to testing.
* Avoid caffeine consumption for 4 h prior to testing and alcohol at least 12 h.
* Maintain normal hydration by drinking to thirst prior to testing.
* Consume a high carbohydrate meal 2 h prior to testing.

Exercise testing

Exercise will be performed in a temperature controlled physiology laboratory. Participants will perform two graded exercise tests, repeated twice. The continuous graded exercise test (CONT) will increase treadmill speed incrementally using three minute stage duration on a motorised treadmill. The initial speed will be individualised designed to evoke a heart rate around 40-50% of one's age predicted maximal heart rate using 206.9 - (0.67* age [yrs]). This will be gauged from a 3 minute low intensity warm-up at the start. The speed will increase by 1 km.hr-1 every three minutes until volitional exhaustion. The gradient of the treadmill will be set at 1 % to reflect energy expenditure of over-ground running. Gradient will only be increased if the performer reaches the limits of their stride frequency and length and therefore it would be inappropriate to continue to increase speed of the belt. The intermittent graded exercise test (INT) will follow the same procedure. However, the speed within each three minute exercise bout will vary every 30 s between the target speed, and a complete pause for 30 s. The acceleration of the treadmill belt will be set to its maximum capability. Participants will be familiarised with this acceleration to ensure safety.

Blood lactate

A post- exercise capillary blood lactate sample will be taken from the participants' finger- tip of their non-dominant hand. The finger -tip will be punctured using a disposable lancet to obtain the capillary blood sample. The small sample of blood is then collected and analysed using a portable blood lactate analyser (Lactate Pro). The finger will be cleaned using an alcohol swab to reduce infection. The researcher taking the blood will be wearing appropriate personal protective equipment including latex-free gloves when obtaining the blood. The blood measure is used as an end-point (among others) to confirm if maximal effort has been performed.

Gas analysis Respiratory data will be recorded continuously throughout each exercise test using an online breath by breath metabolic gas cart (Cortex, metamax). Certified standard calibration gases of 16.4% O2 and 4.5% CO2 will be used (Cryoservice Ltd, Worcester, UK). The turbine flow meter, used for the determination of V ̇E, will be calibrated with a 3 L syringe (Cosmed Srl). Room temperature (°C), relative humidity (%) and barometric pressure (mmHg) will recorded separately from a weather station. Rating of Perceived Exertion (RPE) (modified category-ratio scale) (Foster et al., 2001) expressed as an arbitrary unit (AU) will obtained in the final 15 s of each speed stage.

All breath-by-breath data will be processed using 30 s retrograde averages (Midgley et al., 2007) obtained directly from the metamax software®, with the highest VO2 in the final stages deemed to be VO2max (Midgley et al., 2007). The use of middle 5 of 7 breath averaging will be used for assessment of submaximal data including the ventilatory threshold (Nichols et al 2015). VO2max will be deemed to be achieved if ≥2 of the following criteria are met (Keren et al., 1980): a plateau in VO2 defined as a change of less than 0.2 L.min-1 despite an increasing workload (Howley et al., 1995), a respiratory exchange ratio (RER) of >1.15, a maximal heart rate (HRpeak) within ±10 beats.min-1 of the estimated HRpeak (206.9 - [0.67 x age]), an RPE greater than 8 (Howley et al., 1995) and a 5 min post blood lactate of > 8 mM.

Echocardiography, Electrocardiography and QT interval analysis

A standard transthoracic echocardiogram (TTE) will be used to investigate the existence of any structural cardiac abnormalities. An initial assessment will be performed on the first visit to the laboratory lasting a minimum of 40-45 min. The screening will be carried out by a qualified cardiac physiologist. A 5 minute resting, recovery and exercise 12 lead ECG will be performed using the Mason- Likar set- up. The ECG will be recorded at a paper speed of 25 mm/s. The QT interval will be determined as the interval between the beginning of the Q or R wave to the peak of the T wave, and the point where a tangent drawn along the maximum slope of the descending limb of the T wave crosses the isoelectric TP baseline. The corrected QT interval (QTc) will be calculated using an automated algorithm averaging across 3 beats for each three minute stage, and 60 second recovery phases. We will use a number of different formulas to assess the corrected QT (QTc);

Bazett's (QTc =QT/!RR), Fridericia (QTc=QT/[RR/1000]1/3), Framingham (QTc=QT+[0.154 * {1000-RR}]) Hodges (QTc=QT+1.75 * [{60 000/RR}260])

ELIGIBILITY:
Inclusion Criteria:

* Healthy male soccer players
* Must be participating in ~3 - 6 h of soccer training per week as part of a soccer academy or regional training centre (RTC)

Exclusion Criteria:

* More than one coronary artery disease risk factor
* At least one cardiovascular, respiratory or metabolic disease.
* Have suffered from a lower limb musculoskeletal injury in the past 6 months

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
QT interval duration | Measured during exercise, and immediately following exercise (6 min recovery)
  Duration of the QT interval calculated in each 3 minute stage using various algorithms

SECONDARY OUTCOMES:
Maximal/ Peak Oxygen Uptake | End of exercise (final workload stage) taken as highest value over 30 second average
  Maximum or peak value of oxygen (L/ min) consumed
Ventilatory threshold | During exercise determined using V slope method (10 second, and middle 5 of 7 averages)
  Point during exercise at which ventilation starts to increase at a faster rate than Oxygen consumed

CONTACTS AND LOCATIONS:
Locations (1):
- Sunderland University, Sunderland, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided